CLINICAL TRIAL: NCT01030250
Title: Adjuvant Therapy in Older Versus Younger Women With Breast Cancer: Longitudinal Impact of Adjuvant Chemotherapy on Functional Status, Comorbidity and Quality of Life
Brief Title: Longitudinal Impact of Adjuvant Chemotherapy on Functional Status, Comorbidity and Quality of Life
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08242; R03AG050931 (NIH)
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Adjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Urine to be collected prior to commencement of chemotherapy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Under 65 years: Breast cancer patients receiving adjuvant chemotherapy. Those under 65 years of age will be prospectively evaluated for outcome.
- Over 65 years: Breast cancer patients receiving adjuvant chemotherapy. Those over 65 years of age will be prospectively evaluated for outcome.

SUMMARY:
The goal of this study is to increase our understanding of the adjuvant chemotherapy experience in older and younger adults by prospectively describing the longitudinal trajectory of functional status, comorbidity, and quality of life from before the initiation of chemotherapy to 6 months after the completion of treatment in older (65 and older) and younger (under 65) adults. In addition, we will determine the effect of pre-treatment physical functioning on physical recovery after the course of adjuvant chemotherapy. The secondary objective of this study is to explore if factors other than chronological age (functional status, co-morbid medical conditions, nutritional status, psychological state, cognitive function, and social support) predicts which patients are more likely to experience morbidity (defined as grade 3-5 toxicity, hospitalization, dose reduction or delay, or premature discontinuation of chemotherapy course) from adjuvant chemotherapy.

DETAILED DESCRIPTION:
60% of all cancers and 70% of cancer mortality occur in people greater than 65 years of age, defining cancer as a disease of older adults. Breast cancer is no exception to this rule where almost half of all new breast cancers in the United States are diagnosed in women 65 years of age or older1. Despite the association between cancer and aging, treatment recommendations and data acquired from prospective clinical trials in older women with breast cancer are sparse. As a result, physicians and older adults have limited data to guide treatment recommendation, make dose adjustments and manage toxicities in older adults. Aging is invariably associated with changes in physiology which can impact the pharmacokinetics and pharmacodynamics of cancer therapy. The potential for increased toxic effects in the older patient becomes an important concern. Therefore, it may not be reasonable to extrapolate data regarding toxicity from clinical trials, which primarily include younger, healthier patients. In addition, the age-related impact of adjuvant therapy on the functional status and quality of life of older versus younger adults has not been rigorously evaluated, and risk factors for toxicity, other than chronological age, need to be studied among older adults receiving anthracycline and non-anthracycline based chemotherapy regimens.

The goal of this study is to prospectively describe the longitudinal trajectory of functional status, comorbidity, and quality of life from before the initiation of chemotherapy to 6 months after the completion of treatment in older (65 and older) and younger (under 65) adults. We will determine the effect of pre-treatment physical functioning on physical recovery (ie, physical function at end of chemotherapy and 6 months later) after the course of adjuvant chemotherapy. In addition, we will explore if factors other than chronological age (functional status, comorbid medical conditions, nutritional status, psychological state, cognitive function, and social support) predict which patients are more likely to experience treatment morbidity (defined as grade 3-5 toxicity, hospitalization or urgent care visits, dose reduction or delay, or premature discontinuation of the planned chemotherapy course)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stages I-III breast cancer receiving adjuvant chemotherapy
2. Able to understand English
3. Able to provide informed consent
4. Patients of any age and performance status are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer receiving adjuvant chemotherapy at City of Hope Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2009-06-11 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Describe longitudinal trajectory of physical functional status and quality of life and determine if the patient assessment measure predicts morbidity in adult breast cancer patients from prior to adjuvant chemotherapy to 6 months after end of treatment. | 2 years

SECONDARY OUTCOMES:
Assess potential biomarkers for physiologic age, including Advanced Glycation Endproducts (AGEs) and markers for oxidative stress and inflammation (e.g. 8-OHdG). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arti Hurria, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

REFERENCES:
- [Derived] Yuan Y, Vora N, Sun CL, Li D, Soto-Perez-de-Celis E, Mortimer J, Luu TH, Somlo G, Waisman J, Smith D, Chao J, Katheria V, Synold T, Tran V, Mi S, Levi A, Arsenyan A, Choi J, Zavala L, Yost S, Hurria A. Association of pre-chemotherapy peripheral blood pro-inflammatory and coagulation factors with reduced relative dose intensity in women with breast cancer. Breast Cancer Res. 2017 Aug 29;19(1):101. doi: 10.1186/s13058-017-0895-5. PMID 28851415